CLINICAL TRIAL: NCT05627986
Title: Sensorimotor Cortex Excitability in Shoulder Impingement Syndrome and the Sensorimotor Excitability and Control in Acute/subacute Stage Related to Development of Chronicity
Brief Title: Sensorimotor Cortex Excitability in Shoulder Impingement Syndrome
Status: Completed | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yin-Liang Lin, Assistant Professor, National Yang Ming Chiao Tung University
Other Study IDs: YM111008F
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Shoulder Impingement Syndrome; Chronic Pain; Transcranial Magnetic Stimulation; Electroencephalography; Central Nervous System
Keywords: Shoulder Impingement Syndrome; Corticospinal system; somatosensory system
MeSH Terms: conditions — Shoulder Impingement Syndrome; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- chronic shoulder impingement syndrome: Subjects with shoulder impingement more than 6 months will be included to assess pain threshold, neurophysiological measurements of scapular muscles.
  Interventions: Other: No intervention
- control group: Healthy controls without any shoulder and neck problems will be included to compare the differences in pain threshold, neurophysiological measurements of scapular muscles, scapular kinematics and muscle activation between healthy subjects and subjects with chronic or acute shoulder impingement syndrome.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Shoulder pain is a common musculoskeletal system complaint, accounting for 7-34% of patients in the clinic. The most common shoulder problem is subacromial impingement syndrome (SIS). Up to 45% of individuals with SIS may have unsuccessful treatment and still complain of symptoms after 2 years. This chronicity of pain may not be fully explained by structural injuries or damage, but may be related to sensorimotor changes. Decreased corticospinal excitability and increase inhibition have been found in individuals with SIS. These central motor changes may link to alteration in pain and nociception processing and the somatosensory system, which has been found in individuals with low back pain. Hyperalgesia has been found over both affected and unaffected shoulders in patients with SIS, indicating central and peripheral sensitization. However, no study has investigated whether there are changes in the central somatosensory system. Therefore, the objectives of this proposal are (1) to investigate the corticomotor and somatosensory system in patients with SIS (2) to investigate the relationship between the corticomotor and somatosensory alterations in patients with SIS. Subjects with chronic SIS and healthy subjects were recruited, with 32 people in each group. Electroencephalography (EEG) will be used to collect somatosensory activity, including somatosensory evoked potentials, spectral analysis of EEG oscillations and event-related spectral perturbation (ERSP) of the shoulder movement. Electromyography will be used to record muscle activity. Transcranial magnetic stimulation will be used to test corticomotor excitability, including active motor threshold, motor evoked potentials, cortical silent period, and intracortical inhibition and facilitation. The pressure pain threshold will be collected by a pressure algometer on the muscles of bilateral arms and legs. Pain intensity will be assessed with the Numeric Rating Scale. Shoulder function will be evaluated with the Disability of Arm, Shoulder and Hand questionnaire. Depression will be evaluated with Center for Epidemiologic Studies Depression Scale (CES-D).

ELIGIBILITY:
Inclusion Criteria (chronic impingement syndrome group):

1. individuals have shoulder pain localized at the anterior or lateral aspect of shoulder more than six months
2. are aged 20 to 65 years old
3. shoulder impingement syndrome, which is confirmed by having at least three of the following: (a) positive Neer's test, (b) positive Hawkins-Kennedy test, (c) positive empty can test, (d) positive resisted external rotation test, and (e) presenting painful arc during arm elevation

Inclusion Criteria (acute/subacute impingement syndrome group):

1. individuals have shoulder pain localized at the anterior or lateral aspect of shoulder less than six months
2. are aged 20 to 65 years old
3. shoulder impingement syndrome, which is confirmed by having at least three of the following: (a) positive Neer's test, (b) positive Hawkins-Kennedy test, (c) positive empty can test, (d) positive resisted external rotation test, and (e) presenting painful arc during arm elevation

Inclusion Criteria (health control group)

1. individuals without any shoulder and neck problems
2. sex, age, and hand dominance match to impingement group

Exclusion Criteria:

1. have a history of dislocation, fracture, adhesive capsulities, or surgery of upper extremity
2. arm elevation angle less than 150 degrees
3. a history of direct contact injury to the neck or upper extremities within the past 12 months
4. brain injury and neurological impairment
5. inflammatory cause of the pain (e.g., rheumatoid arthritis)
6. neck pain
7. psychosis and symptom of headache or dizziness
8. allergy to plaster
9. contraindications to the use of TMS, assessed with a safety screening questionnaire

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic impingement syndrome, acute/subacute impingement syndrome and the matched healthy control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Corticomotor excitability measures - Active motor threshold | Immediately during the experiment
  Active motor threshold (AMT) will be described with the percentage (%) of maximum stimulator output (MSO).
Corticomotor excitability measures - Motor evoked potential | Immediately during the experiment
  Motor evoked potential (MEP) will be described with millivolt (mV).
Corticomotor excitability measures - Cortical silent period | Immediately during the experiment
  Cortical silent period (CSP) will be measured with millisecond (ms)
Corticomotor excitability measures - Short interval cortical inhibition | Immediately during the experiment
  Short interval cortical inhibition (SICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Corticomotor excitability measures - Short interval cortical facilitation | Immediately during the experiment
  Short interval cortical facilitation (SICF) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is above 5 ms
Corticomotor excitability measures - Long-interval intracortical inhibition | Immediately during the experiment
  Long-interval intracortical inhibition (LICI) will be defined as percentage (%) of conditioning responses vs testing responses while the inter-stimulus interval is below 5 ms
Corticomotor excitability - Area of cortical mapping | Immediately during the experiment
  Area of cortical mapping will be described with square millimeter (mm2)
Corticomotor excitability - Volume of cortical mapping | Immediately during the experiment
  Volume of cortical mapping will be calculated with multiplying summation of motor evoke potentials on the map (mV) by the area of the map (mm2) with the unit of mV*mm2
Corticomotor excitability - Center of gravity of cortical mapping | Immediately during the experiment
  Center of gravity of cortical mapping will be described in a x-y coordinate system (mm).
Resting brain activity - resting EEG with eye open/closed | Immediately during the experiment
  EEG signals will be processed with power spectrum density analysis to calculate frequency power at Theta (3-8 Hz), alpha (8-13 Hz), beta (13-30 Hz) bands, and Gamma (30 Hz above).
Somatosensory cortical activity - Somatosensory evoked potentials | Immediately during the experiment
  Somatosensory evoked potentials (SEP) will be described with microvolt (µV) and millisecond (ms).
Event-related synchronization or desynchronization - Movement evoked pain potentials | Immediately during the experiment
  Movement evoked pain potentials will be processed with power spectrum density analysis to calculate frequency power at Theta (3-8 Hz), alpha (8-13 Hz), beta (13-30 Hz) bands, and Gamma (30 Hz above) while raising hand.
Muscle activation during arm elevation | Immediately during the experiment
  The root mean square of electromyography (EMG) data of the anterior deltoid and infraspinatus will be normalized by the maximum voluntary contraction amplitude (percentage of maximal voluntary contraction, %) and calculated in two segments, including arm elevating and arm lowering.

SECONDARY OUTCOMES:
Shoulder pain and function-Taiwan version of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Immediately during the experiment
  Subjects will be asked 30 items related to shoulder functional movement. The overall score ranges from 0 (no disability) to 100 (most severe disability).
Depression- Taiwan version of the Center for Epidemiologic Studies Depression Scale (CES-D) | Immediately during the experiment
  Subjects will be asked 20 items to rate how often over the past week they experienced symptoms associated with depression. Response options range from 0 to 3 for each item. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Pressure pain thresholds | Immediately during the experiment
  Pressure pain threshold of bilateral upper trapezius, levator scapulae, infraspinatus, pectoralis major, biceps brachii, middle deltoid and tibialis anterior will each be averaged and will be described with kg/cm2.
Electrical sensory threshold | Immediately during the experiment
  Electrical sensory threshold is the minimal intensity of stimulation required to produce the first perception of sensory and will be described with millivolts (mV).
Electrical pain threshold | Immediately during the experiment
  Electrical pain threshold is the minimal intensity of stimulation required to produce the first perception of pain and will be described with millivolts (mV).

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Liang Lin, PhD, Principal Investigator — National Yang Ming Chaio Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan